CLINICAL TRIAL: NCT06228274
Title: Measurement of the Real Life Efficacy of ARTHRUM 2.5% Health Product Single Injection in Patients Suffering From Knee Osteoarthritis
Brief Title: Assessment of Safety and Efficacy of ARTHRUM 2.5% for Treatment of Painful Osteoarthritis of the Knee
Acronym: ART-ONE75
Status: Completed | Type: Observational
Sponsor: LCA Pharmaceutical (Industry)
Collaborators: BIOSTATEM (Unknown)
Responsible Party: Sponsor
Other Study IDs: 131001
Record Dates: First submitted 2016-07-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic Acid; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARTHRUM 2.5% single injection
  Interventions: Device: ARTHRUM 2.5%

INTERVENTIONS:
Device: ARTHRUM 2.5% — ARTHRUM 2.5%

SUMMARY:
ARTHRUM 2.5% MONO-INJECTION as symptomatic treatment by joint injection extends the conservative therapeutic arsenal in Knee osteoarthritis.

The reduction of functional limits and disabilities induced by knee osteoarthritis as well as improvement of quality of life of patients is a public health need registered amongst the priorities established by the French law of 9 August 2004 relative to Public Health policy. However, the response to this need is not limited to treatment with health products.

This prospective, open, multi-centre trial of the real-life efficacy of ARTHRUM 2.5% aims to demonstrate the efficacy of a single joint injection of this treatment on pain, during 6 months, in the symptomatic treatment of patients suffering from Knee osteoarthritis

DETAILED DESCRIPTION:
Parameters used to determine treatment outcomes include: Western Ontario McMaster Universities Osteoarthritis Index (WOMAC Index), Evaluation of Quality of Life and Handicap and Assessment of therapeutic efficacy

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged over 40
* Suffering from unilateral knee osteoarthritis confirmed radiologically less than six months ago and stage I, II or III according to KELGREEN (knee in extension) and with minimal pain on walking (WOMAC A1) of two points on the LIKERT scale and functional discomfort for at least three months
* Patient able to understand the trial procedure and give his/her consent to take part, in writing
* Patient geographically stable during the trial
* Patient affiliated to the French social security regime or benefiting from such a French regime.

Exclusion Criteria:

* Inflammatory arthritis
* Progressive infectious condition of the knee being studied
* Previous treatment with viscosupplementation for at least one year
* Injection of corticoids into the knee studied for less than three months
* Known hypersensitivity to hyaluronic acid or substances with similar activity
* Anticoagulant treatment in progress
* Insulin-dependent / type I diabetes
* Pregnant or breast-feeding women
* Patient under guardianship or tutorship or under judicial protection
* Patient currently taking part in another clinical research study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Men or women aged over 40
  * Suffering from knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of ARTHRUM 2.5% single joint injection on pain assessed by Likert scale on five levels | 6 months

SECONDARY OUTCOMES:
Safety of ARTHRUM 2.5% under actual conditions of prescription and use: frequency, nature and severity of reported side effects assessed by Likert scale on four levels | 6 months
Reduction of consumption of Analgesics and NSAIDs after ARTHRUM 2.5% intra-articular injection assessed by Likert scale on four levels. | 6 months
Study of ARTHRUM 2.5% intra-articular impact on the Patient's activity assessed by Likert scale on five levels | 6 months
Study of ARTHRUM 2.5% intra-articular impact on the Patient's quality of life by responding one questionnaire assessed by Likert scale on six levels | 6 months
Study of ARTHRUM 2.5% intra-articular impact on the Patient's handicap level by responding one questionnaire assessed by Likert scale on five levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: DOMINIQUE BARON, MD, Study Director — Centre de reeducation et de readaptation fonctionnelles en milieu marin de Trestel

IPD SHARING:
Plan to Share IPD: No